CLINICAL TRIAL: NCT01357993
Title: An Open-Label, Dose-Titration, Long-Term Study to Evaluate the Safety of JNS001 in Adults With Attention-Deficit/Hyperactivity Disorder at Doses of 18 mg, 27 mg, 36 mg, 45 mg, 54 mg, 63 mg or 72 mg Per Day
Brief Title: A Long-Term Study on Safety of JNS001 in Adults With Attention-Deficit Hyperactivity Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR017758; JNS001-JPN-A02 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2011-05-19; First posted 2011-05-23 (Estimated); Last update posted 2014-03-28 (Estimated); Status verified 2014-03

CONDITIONS: Attention-Deficit / Hyperactivity Disorder
Keywords: Methylphenidate hydrochloride; Concerta; Adults; Attention-Deficit / Hyperactivity Disorder; ADHD; Long term safety
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 001 (Experimental): JNS001 18 mg 27 mg and 36 mg tablets (18-72 mg/day) once daily for 48 weeks
  Interventions: Drug: JNS001

INTERVENTIONS:
Drug: JNS001 — 18 mg, 27 mg and 36 mg tablets (18-72 mg/day) once daily for 48 weeks

SUMMARY:
The main purpose of this study is to evaluate long-term safety and tolerability of JNS001 at 18 to 72 mg per day in adults with Attention-Deficit/Hyperactivity Disorder (ADHD).

DETAILED DESCRIPTION:
This is a multicenter, open-label (all people involved know the identity of the intervention), dose-titration (to adjust the dose of a drug until optimal result is reached), long-term safety study in adult patients with a diagnosis of ADHD. The study consists of the Long-term phase (4-week titration period and 44-week maintenance period) and the 1-week Post-study phase. The 4 week-titration period is to find the individualized dose for each patient regardless of the treatments in the preceding study (JNS001-JPN-A01). Patients will be titrated from a starting dose of 18 mg/day for 7 days, and continue with a weekly (+/- 2 days) increment of 9 or 18 mg until an individualized dose is achieved. The titration period will be followed by a 44-week maintenance period which has combined 48-week (1-year) treatment duration with the titration period. During the maintenance period, the dose will be adjusted between 18 to 72 mg depending on the patients' symptoms. In the post-study phase, safety information will be collected after the last dose of the study treatment or premature discontinuation. The study drug will be administered with water once daily in the morning at doses of 18 mg, 27 mg, 36 mg, 45 mg, 54 mg, 63 mg, or 72 mg per day. The study treatment period is 48 weeks (titration period of 4 weeks and maintenance period of 44 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Patients (and their legally-acceptable representative if patients are 18 or 19 years old) must have signed an Informed Consent Form (ICF) indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study
* Patients who completed the preceding study (JNS001-JPN-A01), are considered to be appropriate to continue JNS001 treatment into this extension study by investigator or subinvestigator
* Women of childbearing potential must have a negative urine pregnancy test at the final assessment in the preceding study. If sexually active, continue to use an effective method of birth control throughout the study
* Men must agree to use a double-barrier method of birth control and not donate sperm during the study and for 90 days after receiving the last dose of study drug.

Exclusion Criteria:

* Patients who have reported AEs which would prevent transfer to this study from the preceding study (JNS001-JPN-A01)
* Patients who had been judged ineligible as patients for this study by investigator or subinvestigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2011-05; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) as a Measure of Safety and Tolerability | Throughout the study period (Month 12)

SECONDARY OUTCOMES:
Change in DSM-IV Total ADHD symptoms scores (18 items) of the investigator-rated CAARS-O: SV from baseline of the preceding study (JNS001-JPN-A01) to each visit and to endpoint | Baseline to titration visits (Week 1-4) and to months 2-12 or discontinuation
Change in the scores of the CAARS-S: SV from baseline of the preceding study to each visit and to endpoint | Baseline to months 1-12 or discontinuation
Change in the scores of the CGI-S from baseline of the preceding study in the scores of the CGI-S at each visit and endpoint | Baseline to titration visits (Week 1-4) and to months 2-12 or discontinuation
Change in total score of Q-LES-Q-SF from baseline of the preceding study in the scores of the Q-LES-Q-SFat each visit and endpoint | Baseline to months 1-12 or discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K. Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (29):
- Japan (29):
  - Chiba
  - Chigasaki
  - Chiyoda City
  - Fuchū
  - Fukuoka
  - Fukushima
  - Hamamatsu
  - Higashiosaka
  - Ichikawa
  - Iruma
  - Isehara
  - Kashihara
  - Kishiwada
  - Kobe
  - Kumamoto
  - Kurume
  - Matsuyama
  - Nagasaki
  - Nagoya
  - Nara
  - Neyagawa
  - Osaka
  - Saitama
  - Sakai
  - Sapporo
  - Shibuya City
  - Takatsuki
  - Tokyo
  - Yokohama

REFERENCES:
- See also: An Open-Label, Dose-Titration, Long-Term Study to Evaluate the Safety of JNS001 in Adults with Attention-Deficit/Hyperactivity Disorder at Doses of 18 mg, 27 mg, 36 mg, 45 mg, 54 mg, 63 mg or 72 mg per day — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=1110&filename=CR017758_CSR.pdf